CLINICAL TRIAL: NCT00965549
Title: Comparison of a Basal Plus One Insulin Regimen (Insulin Glargine/Insulin Glulisine) With a Biphasic Insulin Regimen (Insulin Aspart/Insulin Aspart Protamine 30/70) in Type 2 Diabetes Patients Following Basal Insulin Optimisation
Brief Title: Comparison of a Basal Plus One Insulin Regimen With a Biphasic Insulin Regimen in Type 2 Diabetes Patients
Acronym: LanScape
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_04211; 2008-007026-19(EudraCT)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Aspart; insulin glulisine

ARMS (2):
- Lantus + Apidra basal plus one (Experimental): Before randomization (common with arm 2):
  A 1 to 2 weeks of screening period: patients will continue on their current insulin and oral antidiabetic drug (OAD) therapy.
  8 weeks of run-in period: patients will switch their treatment for insulin glargine (one daily injection at bedtime) and all OADs (with the exception of metformin) will be discontinued.
  After randomization:
  24 weeks of treatment period: Insulin (Lantus®) + metformin (if applicable) + a single injection of insulin glulisine (Apidra®), the latter administered at the patients largest meal of the day
  Interventions: Drug: INSULIN GLARGINE (HOE901); Drug: Insulin Glulisine
- NovoMix 30 Biphasic (Active Comparator): Before randomization (common with arm 1):
  A 1 to 2 weeks of screening period: patients will continue on their current insulin and oral antidiabetic drug (OAD) therapy.
  8 weeks of run-in period: patients will switch their treatment for insulin glargine (one daily injection at bedtime) and all OADs (with the exception of metformin) will be discontinued.
  After randomization:
  24 weeks of treatment period: Insulin aspart/ insulin protamine crystallised insulin aspart (NovoMix® 30) + metformin (if applicable)
  Interventions: Drug: Insulin aspart

INTERVENTIONS:
Drug: INSULIN GLARGINE (HOE901) — LANTUS®: Solution for injection. 100U/mL in a prefilled pen (SoloStar®)
  Arms: Lantus + Apidra basal plus one
Drug: Insulin aspart — NovoMix® 30: Suspension for injection. 100U/mL in a prefilled pen (FlexPen®)
  Arms: NovoMix 30 Biphasic
Drug: Insulin Glulisine — APIDRA®: Solution for injection. 100U/mL in a prefilled pen (SoloStar®)
  Arms: Lantus + Apidra basal plus one

SUMMARY:
The primary objective is to demonstrate the non-inferiority at six months of a basal plus one insulin regimen (Lantus plus one injection of Apidra) compared with a biphasic insulin regimen (NovoMix 30) at controlling glycosylated haemoglobin (HbA1c) in type 2 diabetes.

The secondary objective are:

* To compare the proportion of patients in each treatment group reaching HbA1c target (< 7%) at the end of the treatment period
* To compare the rates of hypoglycaemia (total, severe, nocturnal)
* To compare the change in body weight from visit 10 to visit 24
* To compare the change in diabetes specific quality of life and other patient reported outcomes from visit 10 to visit 24

  * Diabetes Treatment Satisfaction Questionnaire - status and change (DTSQs+c)
  * Audit of Diabetes-Dependent Quality of Life (ADDQoL) questionnaire
  * Insulin Treatment Satisfaction Questionnaire (ITSQ)
  * EuroQoL 5 Dimensions (EQ5D) questionnaire
* To record the change in the daily dose of insulin from visit 2 to visit 10 and visit 10 to visit 24

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus
* Patients being treated with Lantus once daily, Levemir once or twice daily or NPH insulin once or twice daily as a single insulin for at least three months 10.0% > or = HbA1c > or = 7.5%
* BMI < or = 40 kg/m²
* If patients are taking oral antidiabetics (OADs), the dose must be stable for at least 1 month
* Ability and willingness to perform blood glucose monitoring using a blood glucose meter and ability and willingness to use a patient diary
* Provision of written informed obtained prior to enrollment in the study

Exclusion criteria:

* Type 1 diabetes mellitus
* Current or previous treatment with an insulin other than basal insulin (biphasic insulin, short acting insulin, rapid-acting insulin analogue)
* Treatment with GLP-1 receptor agonists or with DPPIV inhibitors in the 3 months before screening
* Active proliferative diabetic retinopathy, as defined by the application of photocoagulation or surgery, in the 6 months before screening or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgery during the study (confirmed by an optic fundus exam performed in the 2 years prior to screening)
* Unable or unwilling to enter either of the treatment arms
* Women who are pregnant or lactating (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraceptive method)
* History of hypersensitivity to the study drugs or to drugs with a similar chemical structure
* Treatment with systemic corticosteroids in the 3 months prior to study entry
* Treatment with any investigational product in the 2 months prior to study entry
* Current treatment with any non-selective beta-blockers
* Likelihood of requiring treatment during the study period with drugs not permitted by this clinical protocol
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major disease making implementation of the protocol or interpretation of the study results difficult
* Impaired hepatic function as shown by ALT and/or AST greater than three times the upper limit of normal at screening
* Impaired renal function as shown by serum creatinine >135 µmol/l in men and > 110 µmol/l in women at screening
* History of drug or alcohol abuse
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for follow-up visits, or unlikely to complete the study
* Patient is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Glycosylated Haemoglobin (HbA1c) | At week 7 and week 32

SECONDARY OUTCOMES:
Weight | At week 8 and week 32
Diabetes specific quality of life measured using ADDQoL (Audit of Diabetes-Dependent Quality of Life questionnaire) and other patient reported outcomes measured using EQ5D (EuroQoL 5 Dimensions questionnaire) | Week 8 and week 32
Hypoglycaemia (total, severe and nocturnal) | At week 0 and week 32

CONTACTS AND LOCATIONS:
Overall Officials: Christine van Schalkwyk, MD, Study Director — Sanofi
Locations (74):
- Australia (14):
  - Investigational Site Number 204, Campbelltown
  - Investigational Site Number 205, Campbelltown
  - Investigational Site Number 201, Caulfield
  - Investigational Site Number 210, Daw Park
  - Investigational Site Number 214, Douglas
  - Investigational Site Number 203, Heidelberg
  - Investigational Site Number 206, Herston
  - Investigational Site Number 211, Maroubra
  - Investigational Site Number 207, Meadowbrook
  - Investigational Site Number 212, Melbourne
  - Investigational Site Number 209, Milton
  - Investigational Site Number 213, Nowra
  - Investigational Site Number 202, Parkville
  - Investigational Site Number 208, Southport
- United Kingdom (60):
  - Investigational Site Number 826-109, Aberdeen
  - Investigational Site Number 826-118, Ashton-under-Lyne
  - Investigational Site Number 826-157, Ayr
  - Investigational Site Number 826-149, Barnsley
  - Investigational Site Number 826-135, Bath
  - Investigational Site Number 826-124, Birmingham
  - Investigational Site Number 826-150, Birmingham
  - Investigational Site Number 826-106, Bournemouth
  - Investigational Site Number 826-136, Bradford
  - Investigational Site Number 826-130, Bristol
  - Investigational Site Number 826-114, Bury St Edmunds
  - Investigational Site Number 826-132, Carmarthen
  - Investigational Site Number 826-141, Cheadle
  - Investigational Site Number 826-147, Chester
  - Investigational Site Number 826-112, Chesterfield
  - Investigational Site Number 826-152, Chichester
  - Investigational Site Number 826-159, Cleveleys
  - Investigational Site Number 826-113, Colchester
  - Investigational Site Number 826-119, Cornwall
  - Investigational Site Number 826-162, Crawley
  - Investigational Site Number 826-145, Dafen
  - Investigational Site Number 826-165, Dumfries
  - Investigational Site Number 826-167, Durham
  - Investigational Site Number 826-173, East Kilbride
  - Investigational Site Number 826-105, Edinburgh
  - Investigational Site Number 826-115, Exeter
  - Investigational Site Number 826-160, Fleetwood
  - Investigational Site Number 826-107, Gateshead
  - Investigational Site Number 826-127, Glasgow
  - Investigational Site Number 826-174, Haddington
  - Investigational Site Number 826-164, Hereford
  - Investigational Site Number 826-126, High Wycombe
  - Investigational Site Number 826-102, Hull
  - Investigational Site Number 826-120, Ipswich
  - Investigational Site Number 826-163, Kirkcaldy
  - Investigational Site Number 826-161, Lancaster
  - Investigational Site Number 826-101, Liverpool
  - Investigational Site Number 826-108, Liverpool
  - Investigational Site Number 826-122, Livingston
  - Investigational Site Number 826-110, Llantrisant
  - Investigational Site Number 826-142, London
  - Investigational Site Number 826-123, London
  - Investigational Site Number 826-166, London
  - Investigational Site Number 826-137, Manchester
  - Investigational Site Number 826-156, Mortimer
  - Investigational Site Number 826-140, Newcastle upon Tyne
  - Investigational Site Number 826-138, Newport
  - Investigational Site Number 826-133, Nottingham
  - Investigational Site Number 826-121, Nuneaton
  - Investigational Site Number 826-129, Plymouth
  - Investigational Site Number 826-139, Saint Leonards-on-Sea
  - Investigational Site Number 826-116, Salford
  - Investigational Site Number 826-143, Scunthorpe
  - Investigational Site Number 826-104, Sheffield
  - Investigational Site Number 826-103, St Helens
  - Investigational Site Number 826-111, Stevenage
  - Investigational Site Number 826-131, Stirling
  - Investigational Site Number 826-146, Sunderland
  - Investigational Site Number 826-128, Westbury
  - Investigational Site Number 826-117, York